CLINICAL TRIAL: NCT01292044
Title: The Role of Elastography in the Diagnosis of Thyroid Nodules
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AOI/2010/VT-02; 2010-AO1276-33 (Other: RCB number)
Record Dates: First submitted 2011-02-08; First posted 2011-02-09 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: Thyroid Nodule; Thyroid Neoplasms
Keywords: elastography; cytology
MeSH Terms: conditions — Thyroid Nodule; Thyroid Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- The study population (Experimental): The study population consists of patients for whom an echo-guided fine-needle aspiration was performed for one or more thyroid nodes, and for whom surgical node excision is required.
  Interventions: Other: Elastography

INTERVENTIONS:
Other: Elastography — A conventional thyroid echography performed before a the time of fine needle aspiration will include elastographic measurements for each node under study.

SUMMARY:
The primary objective of this study is to evaluate the role of elastography (along with echographic and cytological data) as a diagnostic tool for thyroid cancer

DETAILED DESCRIPTION:
Ultrasound is considered the first line examination in the exploration of the thyroid nodule. Echotexture analysis often identifies nodules at risk of malignancy, but does not replace or exclude an additional cytological exploration. Cytology, although effective, also has limitations, particularly when samples are vesicular and it is difficult discern between a benign or malignant state. The creation of a noninvasive method in this context could help to avoid invasive tests or "useless" surgical procedures.

Ultrasound elastography, which assesses tissue deformability, may provide valuable information concerning benign soft tissue characteristics, whereas malignant lesions are harder in consistency. Interest in this method, already proposed for other organs, has recently increased due to the emergence of specifically created software that enables objective evaluation of the hardness of the nodule during a conventional ultrasound analysis. The main hypothesis of this study is that elastography should allow better selection of candidates for thyroid surgery.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient is available for six months of follow-up
* The patient is programmed for surgical excision of all nodules determined to be not benign according to cytological criteria

Exclusion Criteria:

* The patient is participating in another study
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* The patient is pregnant
* The patient is breastfeeding
* The patient has a contraindication for a treatment used in this study
* The patient has a contraindication for surgical excision of his/her thyroid nodule
* The patient refused to be operated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2011-11; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
The difference between AUCs for the reference diagnostic method (cytology alone)and the new (cytology + elastography) diagnostic method. | 15 days
  Areas under the curves are estimated using the Wilcoxon-Mann-Chitney statistic. The gold standard is determined by anatomopathological examination of the excised tumor.

CONTACTS AND LOCATIONS:
Overall Officials: Véronique Taillard, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes; Haitham Sharara, MD, Study Director — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, Gard, France